CLINICAL TRIAL: NCT00624416
Title: A Pilot Study: Association of Beta-2 Adrenergic Agonist and Corticosteroid Injection in the Treatment of Lipomas
Brief Title: Association of Beta-2 Adrenergic Agonist and Corticosteroid Injection in the Treatment of Lipomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Lipothera (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 27015
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2012-06-22 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Lipoma
Keywords: Obesity therapy; fat; drug mechanism; adipose tissue; cellular pharmacology
MeSH Terms: conditions — Lipoma; Platelet Glycoprotein IV Deficiency | interventions — Isoproterenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prednisolone and Isoproteronol Together (Other): Beta-adrenergic agonists and corticosteroid
  Interventions: Drug: Prednisolone synthetic cortisone and Isoproterenol together

INTERVENTIONS:
Drug: Prednisolone synthetic cortisone and Isoproterenol together — Approximately 0.2 to 0.4cc of isoproterenol-prednisolone solution (0.04 - 0.08 mg isoproterenol and 0.07 - 0.14 mg prednisolone) in one or more sites in the lipoma depending on its size, 5 days a week for 4 weeks.
  Other Names: Prednisolone combined with Isoproterenol

SUMMARY:
The purpose of this study is to test whether injected medications will increase the amount of fat released by a fat cell. We will compare prednisolone (a synthetic cortisone) combined with isoproterenol (a drug given for asthma) versus using isoproterenol alone. We will also test if injections of isoproterenol and prednisolone will shrink the size of lipomas, which are benign fatty tumors.

DETAILED DESCRIPTION:
Lipomas are benign, non-cancerous fatty tumors that occur under the skin and make a bump that can be easily felt and often seen. The current treatment for lipomas is surgery. Isoproterenol, a medication used for the treatment of asthma and approved for injection under the skin, is known to cause fat cells to give up their fat. The fat cells become resistant to isoproterenol with repeated use. Prednisolone, a synthetic cortisone medication used to treat immune problems like allergy and approved for injection under the skin, keeps the fat cells from becoming resistant to isoproterenol. It is not known, if the fat cells in lipomas act like other fat cells or if the combination of isoproterenol and prednisolone injections would shrink lipomas without surgery. This study is designed to test this possibility.

Subjects will have a screening visit, 2 microdialysis visits a week apart, 20 treatment visits 5 days per week for 4 weeks, and up to 12 follow-up visits a year after treatment visits. During screening, subjects will have a history, physical exam, blood testing, electrocardiogram and a pregnancy testing if female with reproductive capacity. The first microdialysis visit will consist of placing two microdialysis catheters under the skin after the area is numbed. One microdialysis catheter will be in the lipoma and the other under the skin 2 inches away. The microdialysis catheter will connect to a pump, isoproterenol will be infused and the amount of fat breakdown measured. One week later prednisolone will be injected into the lipoma and under the skin 2 inches away. The microdialysis visit will be repeated 24 hours later.

Treatment will consist of injecting the lipoma 5 days a week with a mixture of isoproterenol and prednisolone in the Pennington clinic as a diabetic would inject insulin. Each week the blood pressure, pulse and lipoma will be measured and subjects will be asked how they feel. At the end of the treatment period the physical examination, blood test and electrocardiogram will be repeated.

The insertion of the microdialysis probes under the skin into the fat tissue could be uncomfortable, but numbing medication will be injected first to prevent this problem. At higher doses, isoproterenol could lower blood pressure and increase pulse rate. This should not happen at the doses used, but blood pressure and pulse will be monitored throughout the study. Prednisolone, at higher doses, could decrease the body's production of cortisone. This should not happen at the doses being used, but cortisone in the body will be measured during the trial. Blood tests involve the discomfort of a needle going through the skin of the arm, possible bruising and rarely fainting or infection. Trained technicians and sterile needles will minimize these risks.

ELIGIBILITY:
Inclusion Criteria:

* You are a man or a woman between the ages of 18-60, inclusive.
* You have a body mass index (BMI) between 20 and less than 40 kg/m2. BMI is a number calculated from your height and weight.
* You have a lipoma (a benign fatty tumor) that is 1 inch or more in diameter under the skin of your abdomen or on another area of your body that is easily accessible to study (such as the thigh).
* You have not gained or lost more than 11 pounds in the last 3 months.
* Your exercise routine has been stable for the last 3 months or you are sedentary. Sedentary means you do less than 60 minutes of exercise per week.

Exclusion Criteria:

* You have a history of heart or blood vessel disease.
* Your blood pressure is above 140/90 mmHg.
* You have type 1 diabetes.
* You have a history of kidney or liver disease.
* You have thyroid disease that has not been treated.
* You are a smoker.
* You use a Beta-2 (B2) adrenergic stimulator (a type of drug used to treat asthma), a beta adrenergic blocker (a type of drug used to treat blood pressure) or glucocorticoid medications (a type of drug used to treat immune system disease).
* You have a problem with alcoholism or other substance abuse.
* You are pregnant or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center; Frank Greenway, M.D., Study Director — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisolone and Isoproteronol: Approximately 0.2 to 0.4cc of isoproterenol-prednisolone solution (0.04 - 0.08 mg isoproterenol and 0.07 - 0.14 mg prednisolone) in one or more sites in the lipoma depending on its size, 5 days a week for 4 weeks.
Period: Overall Study
Arm/Group | Prednisolone and Isoproteronol
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prednisolone and Isoproteronol
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Average Percent Volume Reduction in the Lipoma.
Time Frame: Baseline and 4 weeks
Measure: Mean (Full Range); unit: Percent Volume reduction (cc^3)
Units Other Than Participants: Lipoma
Arm/Group | Prednisolone and Isoproteronol
Number analyzed (Participants) | 10
Number analyzed (Lipoma) | 10
Percent Volume reduction (cc^3) | 50 (0.002) [10 to 90]

2. Secondary Outcome: The Number of Lipoma Increased in Volume.
Time Frame: After four weeks of treatment up to one year.
Measure: Number; unit: Lipomas
Units Other Than Participants: Lipoma
Arm/Group | Prednisolone and Isoproteronol
Number analyzed (Participants) | 10
Number analyzed (Lipoma) | 10
Lipomas | 9

3. Secondary Outcome: The Number of Subjects Elected to Have the Lipoma Removed.
Time Frame: After four weeks up to one year.
Measure: Number; unit: participants
Units Other Than Participants: Lipoma
Arm/Group | Prednisolone and Isoproteronol
Number analyzed (Participants) | 10
Number analyzed (Lipoma) | 10
participants | 8

ADVERSE EVENTS:
Arm/Group | Prednisolone and Isoproteronol
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The single case that did not have an increase in lipoma volume showed variability which may have been because of a small lipoma making accurate measurement difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes